CLINICAL TRIAL: NCT05321420
Title: A Randomized Double-blind, Four-Arm Active and Placebo-controlled Dose-Finding Trial to Evaluate the Efficacy, Tolerability, Safety and Dose Response of LYT-100 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: LYT-100 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: ELEVATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PureTech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LYT-100-2022-204
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; lung fibrosis; respiratory disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Respiration Disorders | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo oral administration
  Interventions: Drug: Placebo
- pirfenidone 801 mg TID (Active Comparator): pirfenidone 801 mg TID oral administration
  Interventions: Drug: Pirfenidone
- LYT-100 550 mg TID (Experimental): LYT-100 (Deupirfenidone) 550 mg TID oral administration
  Interventions: Drug: Deupirfenidone
- LYT-100 825 mg TID (Experimental): LYT-100 (Deupirfenidone) 825 mg TID oral administration
  Interventions: Drug: Deupirfenidone

INTERVENTIONS:
Drug: Placebo — placebo
  Arms: Placebo
Drug: Pirfenidone — pirfenidone 801 mg TID
  Arms: pirfenidone 801 mg TID
Drug: Deupirfenidone — Deupirfenidone
  Arms: LYT-100 550 mg TID; LYT-100 825 mg TID

SUMMARY:
This study a randomized, double-blind, four arm study to evaluate the safety and efficacy of LYT-100 compared to pirfenidone or placebo in adults with Idiopathic Pulmonary Fibrosis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, being conducted at centers globally to evaluate the safety and efficacy of LYT-100 compared to pirfenidone or placebo in 240 treatment naïve adult patients with IPF ≥ 40 years in age. Patients will be randomized in a ratio of 1:1:1:1 to receive treatment of LYT-100, pirfenidone, or placebo to be taken daily for up to 183 days (26 week treatment period) with the primary outcome of Rate of decline in Forced Vital Capacity (FVC; in mL) over 26 weeks. Secondary endpoints, including spirometry, inflammatory biomarkers, and patient-reported outcomes will also be evaluated.

After completion of the double-blind period of the study, patients may participate in a long-term extension to evaluate tolerability and long-term safety. Patients receiving LYT-100 in the double-blind period will continue the dose throughout the long-term extension. Patients receiving pirfenidone or placebo in the double-blind period will be re-randomized in a 1:1 ratio to receive LYT-100 550mg or 825mg TID dose throughout the long-term extension.

ELIGIBILITY:
Key Inclusion Criteria:

* Treatment naïve patients or those with <6 months of exposure to nintedanib with physician diagnosed IPF based on ATS/ERS/JRS/ALAT 2018 guidelines
* Idiopathic Pulmonary Fibrosis on HRCT, performed within 12 months of Visit 1 as confirmed by central readers
* DLCO corrected for Hemoglobin (Hb) [visit 1] ≥ 30% and ≤90% of predicted of normal
* FVC ≥ 45% of predicted normal

Key Exclusion Criteria:

* Primary obstructive airway physiology (pre-bronchodilator FEV1/FVC < 0.7 at Visit 1)
* Known explanation for interstitial lung disease, including but not limited to radiation, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans organizing pneumonia, human immunodeficiency virus (HIV), viral hepatitis, and cancer
* Diagnosis of any connective tissue disease, including but not limited to scleroderma/systemic sclerosis, polymyositis/dermatomyositis, systemic lupus erythematosus, and rheumatoid arthritis
* Major extrapulmonary physiological restriction (e.g., chest wall abnormality, large pleural effusion)
* Cardiovascular diseases, any of the following:

  * Uncontrolled hypertension, within 3 months of Visit 1
  * Myocardial infarction within 6 months of Visit 1
  * Unstable cardiac angina within 6 months of Visit 1
* Prior hospitalization for confirmed COVID-19, acute exacerbation of IPF or any lower respiratory tract infection within 3-months of Visit 1

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of decline in Forced Vital Capacity over 26 weeks (Part A) | 26 weeks
  Rate of decline in Forced Vital Capacity (FVC; in mL)

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) percent predicted change (Part A) | Baseline to Week 26
  FVC percent predicted (FVCpp) change from baseline to Week 26
Time to hospitalization or mortality (Part A) | 26 weeks
  Time to hospitalization or mortality due to respiratory cause through 26 weeks
Time to Idiopathic Pulmonary Fibrosis (IPF) progression (Part A) | 26 weeks
  Time to IPF progression through 26 weeks, as defined by a decline in FVC% of 5% or greater or death
Forced Vital Capacity (FVC) percent predicted change (Part B) | 26 Weeks
  FVC percent predicted (FVCpp) change from Week 26 to Week 52
Rate of decline in Forced Vital Capacity over 26 weeks (Part B) | 26 Weeks
  Rate of decline in Forced Vital Capacity (FVC; in mL) from Week 26 to Week 52
Time to Idiopathic Pulmonary Fibrosis (IPF) progression (Part B) | 26 Weeks
  Time to IPF progression from Week 26 to Week 52, as defined by a decline in FVC% of 5% or greater or death

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Graham, MD, Study Director — PureTech
Locations (103):
- United States (22):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Science 37, Los Angeles, California
  - NewportNativeMD, Inc., Newport Beach, California
  - Paradigm Clinical Research Centers, Inc., Redding, California
  - Los Angeles Biomedical Research Institute at Harbor UCLA Medical Center, Torrance, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Accel Research Sites Network, DeLand, Florida
  - Harmony Medical Research Institute, Inc, Hialeah, Florida
  - Piedmont Healthcare, Inc., Atlanta, Georgia
  - Clinical Research Investments, Decatur, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Pulmonix, Greensboro, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Renovatio Clinical - The Woodlands Research Center, The Woodlands, Texas
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - TPMG Clinical Research, Williamsburg, Virginia
- Argentina (14):
  - Instituto Médico de la Fundación de Estudios Clinicos / Fundación Estudios, Rosario, Santa Fe Province
  - Aprillus Asistencia e Investigación, Buenos Aires
  - CEMER Centro Medico de Enfermedades Respiratorias, Buenos Aires
  - Instituto de Medicina Respiratoria - IMER, Córdoba
  - Respira Salud Clinica Integral, Godoy Cruz
  - Instituto Ave Pulmo - Fundacion Enfisema, Mar del Plata
  - Polo de Salud Vistalba, Mendoza
  - CIMRO- Centro de Investigación Médica Respiratoria Oncológica, Mendoza
  - INSARES - Instituto de Salud Respiratoria, Mendoza
  - Centro Médico Dharma, Mendoza
  - Instituto de Enfermedades Respiratorias e Investigación Clínica, San Juan Bautista
  - Investigaciones en Patologías Respiratorias, San Miguel de Tucumán
  - Instituto del Buen Aire, Santa Fe
  - Clinica Central S.A., Villa Regina
- Chile (4):
  - Clinica Maule, Maule
  - Centro de Estudios Clinicos, Santiago
  - Clinica Universidad de Los Andes, Santiago
  - Centro Respiratorio Integral, Valparaíso
- Colombia (3):
  - Fundacion Cardiomet CEQUIN, Armenia
  - Instituto Neumologico del Oriente S.A., Bucaramanga
  - Centro de Investigaciones Clinicas S.A.S, Cali
- Georgia (5):
  - National Ceneter for Tuberculosis and Lung Diseases JSC, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic LLC, Tbilisi
  - Emergency Cardiology Center by Academician G. Chapidze LLC, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD The First Medical Center, Tbilisi
- Greece (6):
  - University Hospital Alexandroupolis, Alexandroupoli
  - "Sotiria" Chest Diseases Hospital of Athens, Athens
  - University General Hospital "Attikon", Athens
  - Athens Medical Center, Athens
  - University General Hospital of Patras, Pátrai
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- India (10):
  - Rhythm Heart Institute Vadodara, Vadodara, Gujarat
  - Sparsh Super Specialty Hospital, Bengaluru, Karnataka
  - Mgm Medical College And Hospital, Aurangabad, Aurangabad, Maharashtra
  - Government Medical College and Hospital Aurangabad, Aurangabad, Maharashtra
  - Oriion Citicare Super Specialty Hospital, Aurangabad, Maharashtra
  - Getwell Hospital and Research Institute, Nagpur, Maharashtra
  - Govt. General and Chest Hospital, Hyderabad, Telangana
  - Apollo Spectra Hospital, Kanpur, Uttar Pradesh
  - Nil Ratan Sircar Medical College And Hospital, Kolkata, Kolkata, West Bengal
  - BHS Lakeview Heart, Belagāve
- Malaysia (6):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Pulau Pinang, George Town
  - Hospital Serdang, Kajang
  - Institut Perubatan Respiratori, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
- Mexico (5):
  - Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León
  - Integral Health Medical Unit, San Nicolás de los Garza, Nuevo León
  - CALPULAB, Calpulalpan
  - Oaxaca Site Management Organization, Oaxaca City
  - ONCARE Group, San Pedro Garza García
- Philippines (3):
  - St. Luke's Medical Center - Global City, City of Taguig
  - Philippine General Hospital, Manila
  - Lung Center of the Philippines, Quezon City
- Romania (3):
  - S.C. Netconsult SRL, Iași
  - S.C. Lavinia Davidescu Clinic SRL, Oradea
  - "Dr. Victor Babes" Clinical Hospital of Infectious Diseases and Pneumophtisiology, Timișoara
- South Africa (5):
  - Durban Lung Centre, Durban
  - WITS Clinical Research, Johannesburg
  - Ahmed Kathrada Lenmed Private Hospital, Johannesburg
  - Netcare Milpark Hospital, Parktown
  - Ryexo Clinical Research, Pretoria
- South Korea (13):
  - The Catholic University Of Korea Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Hanyang University - Myongji Hospital, Goyang-si, Gyeonggi-do
  - InJe University Haeundae Paik Hospital, Busan
  - Keimyung University - Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - CHA Bundang Medical Center, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Thailand (4):
  - Siriraj Hospital, Bangkok
  - Khon Kaen University, Khon Kaen
  - Central Chest Institute Of Thailand, Nonthaburi
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Recruiting website for patients in the United States — http://www.elevateipf.com